CLINICAL TRIAL: NCT02925650
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamic (PD) Effects of Posiphen® in Subjects With Early Alzheimer's Disease (AD)
Brief Title: Safety, Tolerability, PK and PD of Posiphen® in Subjects With Early Alzheimer's Disease
Acronym: DISCOVER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QR15001; ADC-042-DISC (Other: Alzheimer's Disease Cooperative Study (ADCS))
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; SILK™; Pharmacodynamics; Safety; Pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease | interventions — phenserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): The study drug Posiphen dosage of 60mg is to be taken orally in divided doses, three times per day for a total 23-25 days.
  Interventions: Drug: Posiphen
- Medium Dose (Experimental): The study drug Posiphen dosage of 120mg is to be taken orally in divided doses, three times per day for a total 23-25 days.
  Interventions: Drug: Posiphen
- High Dose (Experimental): The study drug Posiphen dosage of 180mg is to be taken orally in divided doses, three times per day for a total 23-25 days.
  Interventions: Drug: Posiphen
- Placebo (Placebo Comparator): The Placebo comparator is to be taken orally in divided doses, three times per day for a total 23-25 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Posiphen — oral solid dosage form capsule
  Arms: High Dose; Low Dose; Medium Dose
Drug: Placebo — oral solid dosage form capsule
  Arms: Placebo

SUMMARY:
This study evaluates the safety and pharmacological effects of 3 different doses of Posiphen® when compared to a placebo, in adult male and female patients with early Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Posiphen®, which was discovered by the US National Institute on Aging (NIA) is a small, orally active, experimental drug that specifically inhibits the synthesis of amyloid precursor protein (APP), Tau and α-Synuclein. It is distinct from other Alzheimer's disease drugs currently in development, because it inhibits the formation of several toxic proteins, rather than removing individual toxic protein after they are produced. Posiphen has potential utility as a disease modifying treatment for AD. The present study will confirm the pharmacokinetics (PK) of Posiphen and its metabolites in plasma and cerebral spinal fluid (CSF). It will also measure the effects of a 23-25 day treatment period with Posiphen on the CSF and plasma levels of a number of biomarkers, inflammatory factors and control proteins. It will also expand the safety data in humans by extending the treatment period from 10 days to a treatment period from 23-25 days. In addition, this study will measure concentrations of various soluble biomarkers in CSF and use the SILK™ assay methods to directly measure the effect of Posiphen on the fractional synthesis rate of Aβ40 in CSF, which will help guide the further development of Posiphen and determine the feasibility of SILK™ in a multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 55 to 89 years (inclusive), in good health, no frailty.
2. Female participants must be post-menopausal for at least 2 consecutive years or surgically sterile (bilateral tubal ligation, hysterectomy or bilateral oophorectomy) for at least 6 months prior to screening.
3. Female participants will be given a urine pregnancy test at the screening visit for which they should test negative.
4. Clinical profile consistent with MCI or mild AD, consistent with the core clinical criteria outlined in the NIA-AA Guidelines (2011).
5. MMSE score between 17 and 30 (inclusive).
6. CDR global score of 0.5 with a memory score of 0.5 or greater, or CDR global score of 1.0.
7. Participant likely to tolerate all study procedures per PI judgment.
8. To qualify for entry, subjects will have a CSF Abeta42-Abeta40 ratio below 0.131 that is consistent with Alzheimers disease as measured via mass spectrometry by C2N.
9. General cognition and functional performance sufficiently preserved that the subject can provide written informed consent.
10. A minimum of 6 years of education or good work history.
11. Study partner is available who has frequent contact with the subject (e.g., average of 10 hours per week or more), and can accompany the subject to most visits to answer questions about the subject. The study partner is required to attend the entire screening visit and the baseline visit. The study drug is dispensed to the participant at the baseline visit and the study partner (or other individual) should also oversee study drug administration if needed to ensure compliance with dose regimen. At a minimum, the study partner should stay for the first 3 hours of the confinement visit and return at the discharge to drive the subject home.
12. No evidence of current suicidal ideation or previous suicide attempt in the past month as evaluated in the Columbia Suicide Severity Rating Scale.
13. MRI scan within the 12 months prior to screening without evidence of infection, infarction, or other focal lesions and without clinical symptoms suggestive of intervening neurological disease. Lacunes that are not believed to contribute to the subjects cognitive impairment are permissible. If there is no MRI available within a 12-month timeframe, then an MRI must be performed as part of the screening procedures for eligibility.
14. Stability of permitted medications for 4 weeks prior to baseline. NOTE: Cholinesterase inhibitors and or memantine are allowable only if stable for 12 weeks prior to screen. If taking Arciept (donezepil), no more than 10 mg/day is permitted during the course of the study.
15. Adequate visual and hearing ability (physical ability to perform all the study assessments).
16. Good general health with no disease expected to interfere with the study. Subjects may have common age-related disorders (i.e., hypertension, type II diabetes, dyslipidemia, and hypothyroidism) as long as these disorders are being controlled by diet or medication.
17. Must speak English, Spanish, or Korean fluently.

Exclusion Criteria:

1. Has a history of a psychiatric disorder such as schizophrenia, bipolar disorder or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM). Mild depression or history of depression that is stable on treatment with a tricyclic antidepressant SSRI or SNRI medication at a stable dose is acceptable.
2. Other neurodegenerative diseases, including Parkinsons disease and Huntingtons disease, or cerebral tumor.
3. Dementia other than AD, such as Acquired Immunodeficiency Syndrome (AIDS), Creutzfeldt-Jakob disease (CJD), Lewy Bodies dementia (LBD), Cerebrovascular dementia (CVD), Progressive Supranuclear Palsy (PSP), or normal pressure hydrocephalus (NPH).
4. History of a seizure disorder.
5. Clinically significant abnormalities in screening laboratory or ECG results.
6. Has current serious or unstable illness including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease or other conditions that, in the investigators opinion, makes them ineligible for participation in this study.
7. Has four or more microinfarcts as noted in the MRI scan.
8. Has cancer or has had a malignant tumor within the past 3 years, except patients who underwent potentially curative therapy with no evidence of recurrence. (Patients with stable untreated prostate cancer or skin cancers are not excluded).
9. According to the criteria of the most current version of the DSM, alcohol abuse, alcohol dependence, or drug abuse in the past 5 years.
10. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 16 weeks prior to screening. (The end of a previous investigational trial is the date the last dose of an investigational agent was taken).
11. Resides in a skilled nursing facility.
12. Subjects with infection or inflammation of the skin or skin disease at or in proximity to the lumbar puncture site.
13. History of lumbar spine surgery or chronic low back pain (CLBP).
14. Subjects whom the site PI deems to be otherwise ineligible.
15. Has a deep brain stimulator (DBS).

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSD Alzheimer's Disease Research Center, La Jolla, California
  - IU Health Partners, Adult Neurology Clinic, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University Sleep Medicine Center, Brentwood, Missouri
  - Columbia University Medical Center Sergievsky Center Taub Institute, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data from this research will be shared with other researchers pursuant to the 02/26/2003 "NIH Final Statement on Sharing Research Data". The ADCS through its Data and Sample Sharing Committee (DSSC) will receive requests for sample and data sharing. The ADCS grants access to de-identified data to qualified scientists who complete the request process and agree to conditions in an ADCS/UCSD Data Use Agreement (DUA) and the ADCS Publications Policy. After approval and receipt of the fully executed DUA, applicants are authorized to acquire data. Non-compliance with the DUA, including the requirement to provide requested updates will jeopardize further access to data. The same process and Committee reviews and approves biosample requests. If a request for biosample sharing is approved, a Material Transfer Agreement (MTA) will be negotiated between UCSD/ADCS and the requesting researcher or organization.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01 August 2023
Access Criteria: Data requestors must complete an ADCS Data and Sample Sharing request form which will be reviewed by the ADCS DSSC. Upon approval, requestors must complete a Data Use Agreement (DUA) prior to accessing the data.
URL: https://www.adcs.org/data-sharing/

REFERENCES:
- [Derived] Galasko D, Farlow MR, Lucey BP, Honig LS, Elbert D, Bateman R, Momper J, Thomas RG, Rissman RA, Pa J, Aslanyan V, Balasubramanian A, West T, Maccecchini M, Feldman HH. A multicenter, randomized, double-blind, placebo-controlled ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) effects of Posiphen in subjects with early Alzheimer's Disease. Alzheimers Res Ther. 2024 Jul 5;16(1):151. doi: 10.1186/s13195-024-01490-z. PMID 38970127
- [Derived] Galasko D, Farlow MR, Lucey BP, Honig LS, Elbert D, Bateman R, Momper J, Thomas R, Rissman RA, Pa J, Aslanyan V, Balasubramanian A, West T, Maccecchini M, Feldman HH. A multicenter, randomized, double-blind, placebo-controlled ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) effects of Posiphen in subjects with Early Alzheimer's Disease. medRxiv [Preprint]. 2024 Mar 22:2024.03.20.24304638. doi: 10.1101/2024.03.20.24304638. PMID 38562783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
Started | 5 | 5 | 1 | 7
Completed | 4 | 5 | 1 | 5
Not Completed | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 1 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 1 | 5
  >=65 years | 4 | 3 | 0 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 0 | 3 | 8
  Male | 0 | 5 | 1 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 5 | 1 | 6 | 17
  Unknown, Not Reported | 0 | 0 | 0 | 1 | 1
  Not-Hispanic or Latino | 5 | 5 | 1 | 6 | 17
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 1 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Multiple Ascending Doses of Posiphen: Reports of Adverse Events or Study Discontinuations
Description: Number of adverse events or study discontinuations, broken down by dose arm (i.e. Low vs. Medium vs. High vs. Placebo), and further broken down by relatedness to Posiphen (Definitely Related, Probably Related, Possibly Related, Unlikely Related, Unrelated)
Time Frame: Up to 25 days
Measure: Number; unit: events
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
Number analyzed (Participants) | 5 | 5 | 1 | 7
events
  Definitely Related | 0 | 0 | 0 | 0
  Probably Related | 0 | 1 | 0 | 0
  Possibly Related | 1 | 0 | 0 | 2
  Unlikely Related | 2 | 3 | 0 | 2
  Unrelated | 9 | 11 | 0 | 6
  Total | 12 | 15 | 0 | 10

2. Primary Outcome: The Levels of Posiphen and Its Metabolites Will be Determined in Plasma
Description: Mean plasma concentrations of levels of posiphen tartrate, N1 desmethyl posiphen, and N8 desmethyl Posiphen metabolite were determined for each of the three dose cohorts (Low Dose, Medium Dose, High Dose) by a protein precipitation extraction method using a high performance liquid chromatographic mass spectrometric detection method, with a linear weighted regression to determine their concentrations.
Time Frame: The confinement visit occurred following 21-23 days of treatment with either Posiphen or placebo, while also allowing a +/- 2-day visit window. Plasma was collected at 0, 2, 4, 8, 12, 16, 20, and 24hrs during the confinement visit.
Population: Participants in the Placebo Arm/Group were not given study drug. Therefore, measurements of study drug, Posiphen, and its metabolites were not performed on the Placebo Arm/Group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 5 | 5 | 1
ng/mL
  Posiphen | 7.16 (4.25) | 9.51 (5.77) | 12.01 (0)
  N1 metabolite | 1.29 (0.77) | 3.02 (1.4) | 2.51 (0)
  N8 metabolite | 2.25 (1.36) | 5.04 (1.8) | 3.35 (0)

3. Primary Outcome: The Levels of Posiphen and Its Metabolites Will be Determined in Cerebrospinal Fluid (CSF)
Description: Mean CSF concentrations of levels of posiphen tartrate, N1 desmethyl posiphen, and N8 desmethyl Posiphen metabolite were determined for each of the three dose cohorts (Low Dose, Medium Dose, High Dose) by a protein precipitation extraction method using a high performance liquid chromatographic mass spectrometric detection method, with a linear weighted regression to determine the concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 5 | 5 | 1
ng/mL
  Posiphen | 0.46 (0.3) | 0.73 (0.52) | 0.71 (0)
  N1 metabolite | 0.02 (0.04) | 0.28 (0.3) | 0 (0)
  N8 metabolite | 0.35 (0.26) | 0.77 (0.43) | 0.15 (0)

4. Primary Outcome: Fractional Synthesis Rate of Aβ40 in CSF Using the SILK™ Technique With Multiple Doses of Posiphen
Description: The fractional synthesis rate (FSR) of Aβ40 was measured in the CSF using the SILK™ technique. FSR is a measure of the rate of Aβ synthesis in the brain. During 13C6-leucine infusion, 13C6-leucine is incorporated into newly synthesized proteins throughout the body, including the brain, in proportion to the available 13C6-leucine. This FSR is calculated as the rate of change of the ratio of 13C6-leucine-labeled Aβ proteins to unlabeled Aβ proteins in the lumbar CSF between 6 to 16 hours, normalized to the ratio of labeled to unlabeled leucine amino acid in plasma. It is reported as a fraction of 13C6-leucine-labeled to unlabeled Aβ proteins per hour. The ratio of Aβ in CSF containing 13C6-leucine to that containing unlabeled leucine is measured using mass spectrometry.
Time Frame: The confinement visit occurred following 21-23 days of treatment with either Posiphen or placebo, while also allowing a +/- 2-day visit window. CSF was collected between 6 and 16hrs during the confinement visit.
Population: 15 participants completed the Confinement visit and had sufficient samples to enable this analysis
Measure: Mean (Full Range); unit: fraction labeled:unlabeled Aβ40 per hr
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
Number analyzed (Participants) | 4 | 5 | 1 | 5
fraction labeled:unlabeled Aβ40 per hr | 0.0405 [0.0298 to 0.0431] | 0.0400 [0.0373 to 0.0511] | 0.0206 [0.0206 to 0.0206] | 0.0375 [0.0319 to 0.0449]

5. Secondary Outcome: Feasibility of CSF Catheter Study With SILK™ Technology to Evaluate Rates of Enrollment
Description: Feasibility of CSF Catheter Study with SILK™ Technology was determined by comparing the total number of participants enrolled, randomized and treated with study drug in the trial to the total number of participants who completed the CSF Catheter Study across all participating sites.
Time Frame: Up to 25 days
Population: Overall number of participants completing the protocol
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment Arms: Participants who were randomized to receive Active Treatment (Posiphen 60mg, 120mg or 180mg)
- Placebo Arm: Participants who were randomized to receive Placebo
Arm/Group | Active Treatment Arms | Placebo Arm
Number analyzed (Participants) | 11 | 7
Participants | 10 | 5

6. Secondary Outcome: Feasibility of CSF Catheter Study With SILK™ Technology to Evaluate %CSF Samples With Enough Volume for Testing
Description: The % of cerebrospinal fluid samples with sufficient volume for testing will be determined across study participants during the SILK sampling procedure
Time Frame: Up to 25 days
Population: The % of CSF samples with sufficient volume for testing will be determined across study participants during the SILK sampling procedure
Measure: Number; unit: percentage of CSF samples
Groups:
- All Randomized Participants Who Completed 36 Hour Confinement Visit (n=15): Time points where sufficient CSF samples (6 ml) were collected across 285 time points (15 participants * 19 CSF collection time points).
Arm/Group | All Randomized Participants Who Completed 36 Hour Confinement Visit (n=15)
Number analyzed (Participants) | 15
percentage of CSF samples | 81.75

7. Secondary Outcome: Feasibility of CSF Catheter Study With SILK™ Technology to Evaluate Research Satisfaction
Description: Research satisfaction will be evaluated by qualitative response to 14 questions asked to participants about their experience with the study procedures. Responses will be grouped and reported by common themes
Time Frame: Up to 25 days
Measure: Number; unit: percentage of participants
Groups:
- All Randomized Participants: Responses to 14 questions from Research Satisfaction Survey (RSS) from all randomized participants
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 15
percentage of participants
  Rated "Excellent" for quality of tests and attention received during participation in the study. | 94
  Reported "Almost all of my expectations have been met" by the research program. | 81
  Reported "Yes, definitely" they would recommend this research program to a friend. | 94
  Reported "Yes, definitely" they would choose to participate again. | 87.5
  Reported "Volunteering" as what they liked best about the study. | 31
  Reported "Time Commitment" as what they liked least about the study. | 31
  Reported "Yes", the 36 hour catheter procedure was done. | 100
  Reported "No" adverse events were associated with the 36hr catheter procedure. | 73
  Reported "Excellent" as the quality of the 36hr catheter procedure and attention they received. | 80
  Reported the catheter procedure was "almost all of what I expected." | 67
  Reported they liked best was "participating in cutting edge research and interacting with the team". | 100
  Reported "Other" as what they liked least about the 36hr catheter procedure. | 47
  Reported "Other" as what they would change about the 36hr catheter procedure. | 71
  Reported they would change the number of visits. | 50

8. Secondary Outcome: Pharmacodynamic and PK-PD Effects on CSF Alzheimer's Disease Biomarkers
Description: Aβ38, Aβ40, Aβ42, sAPPα, sAPPβ, and T-Tau were sampled at Screening and at the start of the confinement visit. Results of these measures were reported as a least square means, calculated as the change between the measured values at the start of the confinement visit and Screening in ng/mL.
Time Frame: CSF was sampled at Screening and at the start of the confinement visit, which occurred following 21-23 days of treatment with either Posiphen or placebo, while also allowing a +/- 2-day visit window.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Active Treatment Arms | Placebo Arm
Number analyzed (Participants) | 10 | 7
ng/mL
  Aβ38 | 0.391 (0.173) | 0.593 (0.199)
  Aβ40 | 1.73 (0.998) | 3.13 (1.151)
  Aβ42 | 0.107 (0.0653) | 0.211 (0.0753)
  sAPPα | 6.49 (5.75) | -3.5 (9.07)
  sAPPβ | 19.1 (16.8) | -28.6 (26.5)
  Total Tau | 186.4 (79.1) | 53.7 (124.9)

9. Secondary Outcome: Assessment of Mental Status Effects
Description: The short-term effects of Posiphen on mental status will be measured using the Mini-Mental State Examination (MMSE). The MMSE is a brief, global cognitive measure that includes orientation, memory, attention, concentration, naming, writing, repetition, comprehension, and construction. The total score ranges from 0 (worst) to 30 (best performance). Results of the MMSE for this trial were reported as a raw change score, calculated as the change between the total scores at two evaluation time points (Baseline, Pre-Confinement Visit) and where negative values are worse and positive values are better.
Time Frame: MMSE was administered at Baseline and at the Pre-Confinement Visit 1-3 days prior to the Confinement Visit. This confinement visit occurred following 21-23 days of treatment with either Posiphen or placebo, while also allowing a +/- 2-day visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
Number analyzed (Participants) | 5 | 5 | 1 | 7
score on a scale | -1.4 (0.89) | 1.2 (2.39) | -1 (0) | 1.14 (2.12)

10. Secondary Outcome: Assessment of Neuropsychiatric Effects
Description: The Neuropsychiatric Inventory (NPI) was used to measure the frequency and severity of neuropsychiatric symptoms. On this scale frequency ratings range from 0 (no symptoms) to 4 (very frequently, once or more per day or continuously). Severity ratings range from 0 (no severity) to 3 (severe). The score for each of 12 symptoms measured in the scale is the product of severity and frequency within that symptom. The total score for the NPI is the sum of all 12 symptom item scores, for a highest possible total score of 144 in individuals with maximal symptoms, and a lowest possible total score of zero (0) in fully asymptomatic individuals. Lower scores are better and higher scores indicate more neuropsychiatric symptoms. Results are calculated as the change between the total scores at two evaluation time points (Baseline, Pre-Confinement Visit) with negative scores being better and positive scores being worse.
Time Frame: NPI was administered at Baseline and at the Pre-Confinement Visit 1-3 days prior to the Confinement Visit. This confinement visit occurred following 21-23 days of treatment with either Posiphen or placebo, while also allowing a +/- 2-day visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
Number analyzed (Participants) | 5 | 5 | 1 | 7
score on a scale | -2.6 (2.88) | 3.4 (8.47) | -9 (0) | -3.86 (8.09)

11. Secondary Outcome: Assessment of Cognitive Effects
Description: The short-term effects of Posiphen on cognition were measured using the The Alzheimer's Disease Assessment Scale-Cognitive 12 (ADAS-Cog12). The ADAS-Cog is a structured scale that evaluates memory (word recall, word recognition), reasoning, language (naming, comprehension), orientation, ideational praxis and constructional praxis. The test is scored in terms of errors, with higher scores reflecting poorer performance and greater impairment. Total ADAS-Cog12 scores can range from 0 to 80, with lower scores being better and higher scores being worse. Results of the ADAS-Cog12 for this trial are reported as a raw change score, calculated as the change between the total scores at two evaluation time points (Baseline, Pre-Confinement Visit) with negative scores being better and positive scores being worse.
Time Frame: ADAS-Cog12 was administered at Baseline and at the Pre-Confinement Visit 1-3 days prior to the Confinement Visit. This confinement visit occurred following 21-23 days of treatment with either Posiphen or placebo, also allowing a +/- 2-day visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment Arms | Placebo Arm
Number analyzed (Participants) | 11 | 7
score on a scale | -0.55 (6.04) | -1.57 (5.19)

ADVERSE EVENTS:
Time Frame: From Randomization through Study Day 25.
Arm/Group | Low Dose | Medium Dose | High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 0/1 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=5) | Medium Dose (N=5) | High Dose (N=1) | Placebo (N=7)
agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
catheter site swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
fatigue (General disorders) | 1 | 0 | 0 | 0
headache (Nervous system disorders) | 1 | 2 | 0 | 3
injection site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
injection site swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
lethargy (General disorders) | 0 | 1 | 0 | 0
medical device complication (Gastrointestinal disorders) | 0 | 2 | 0 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
pain (General disorders) | 0 | 0 | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
traumatic lumbar puncture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
tremor (Nervous system disorders) | 0 | 0 | 0 | 2
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT02925650/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT02925650/SAP_001.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT02925650/ICF_003.pdf